CLINICAL TRIAL: NCT04805983
Title: An Open-Label, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Receptor Occupancy of BMS-984923
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics and Receptor Occupancy of BMS-984923
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Adam Mecca, Assistant Professor of Psychiatry; Associate Director, Alzheimer's Disease Research Unit; Faculty, Alzheimer's Disease Research Center (ADRC), Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000028864; 1U01AG058608-01A1 (NIH)
Record Dates: First submitted 2021-03-14; First posted 2021-03-18 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The study will enroll four cohorts of 6 participants each. Study drug will be administered in sequentially increasing dose groups. For all 6 participants at a dose cohort, a safety assessment review will be completed prior to advancing the next higher dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 10 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923
- 40 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923
- 70 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923
- 100 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923
- 150 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923
- 200 mg BMS-984923 (Experimental)
  Interventions: Drug: BMS-984923

INTERVENTIONS:
Drug: BMS-984923 — Day 1: Admission, administration of study drug, and 2 night in-patient stay; Day 3: Discharge following the completion of all scheduled procedures.

SUMMARY:
This project seeks to develop a novel disease-modifying compound for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety, tolerability, and pharmacokinetics of BMS-984923 in healthy participants. A secondary objective of this study is to conduct a receptor occupancy sub-study aimed at determining drug receptor occupancy at each dose using [18F]FPEB Positron Emission Tomography.

ELIGIBILITY:
Inclusion Criteria:

* No history of cognitive impairment
* Capable of providing written informed consent and willing to comply with all study requirements and procedures
* Participant is not pregnant, lactating, or of childbearing potential

  1. Non-childbearing potential for women is defined as postmenopausal (last natural menses greater than 24 months; menopausal status will be documented with serum follicle stimulating hormone (FSH) or documentation of bilateral tubal ligation or hysterectomy
  2. Male participants who are sexually active with a woman of child-bearing potential must agree to use condoms during the trial and for 3 months after the last dose unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
  3. Male participants must also agree not to donate sperm for 90 days after the last dose. -
* Glasgow Coma Scale Score of 15 (97)
* Clinical Dementia Rating Score of 0 (93)
* Has a reliable study partner who has frequent contact with the participant (e.g., average of 10 hours per week or more), who can be available for study partner assessments, who can accompany the participant for 48 hours, without absence, after discharge from Visit 2.

Score on the Mini Mental Status Exam > 26 (95)

* Objective memory scores within normal range for age evidenced by a score no more than 1.5 standard deviations below the education adjusted cutoff on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (the maximum score is 25).

  1. >8 for 16 or more years of education
  2. >4 for 8-15 years of education
  3. >2 for 0-7 years of education

Receptor Occupancy Substudy Eligibility Criteria

* Eligibility for and enrollment in Main Study
* Participant consent to the optional substudy

Exclusion Criteria:

* Body mass index (BMI) ≥ 35 kg/m2 or body weight < 50 kg.
* Significant cerebrovascular disease: Modified Hachinski score > 4.
* Any significant neurologic disease, such as AD, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
* Major depression, bipolar disorder as described in DSM-IV within the past 1 year.
* Psychotic features, agitation or behavioral problems within 3 months, which could lead to difficulty complying with the protocol.
* History of schizophrenia (DSM IV criteria).
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
* Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results, or the patient's ability to participate in the study.
* Clinically significant abnormalities in B12 or Thyroid Function Tests that might interfere with the study.

Use of psychoactive medications (typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.

* Use of medications with significant CYP1A2, 2D6, or 3A4 inhibitor or inducer activity (See appendix for a list of these medications) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
* Use of anticoagulants within 30 days or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
* Use of investigational amyloid lowering therapies within 2 months prior to study drug administration and for the duration of the trial.
* Use of another investigational agent within 30 days or 5 half-lives (whichever is greater) prior to screening and for the duration of the trial.
* Neutropenia defined as absolute neutrophils count of < 1,500/microliter.
* Thrombocytopenia defined as platelet count < 100,000/microliter.
* Clinically significant abnormalities in screening laboratories, including Aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN); Alanine aminotransferase (ALT) >1.5 times ULN; Total bilirubin >1.5 times ULN; Serum creatinine >2.0 times ULN.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mecca, MD, PhD, Principal Investigator — Assistant Professor of Psychiatry; Associate Director, Alzheimer's Disease Research Unit; Faculty, Alzheimer's Disease Research Center (ADRC)
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed Baseline (Study Day 1) | 6 | 6 | 6 | 6 | 6 | 6
Completed Inpatient Treatment (Study Day 3) | 6 | 6 | 6 | 6 | 6 | 6
Completed In-Clinic Follow-Up (Study Day 4) | 6 | 6 | 6 | 6 | 6 | 6
Completed Phone Visit Follow-Up (Study Day 5) | 6 | 6 | 6 | 6 | 6 | 6
Completed In-Clinic Final Follow- Up/Completed Protocol (Study Day 7) | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (3.2) | 71.3 (5.6) | 70.3 (2.5) | 68.3 (3.5) | 72.8 (6.1) | 68.1 (9.1) | 70.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 3 | 2 | 21
  Male | 2 | 2 | 2 | 2 | 3 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 4 | 5 | 6 | 6 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 6 | 6 | 5 | 6 | 6 | 6 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 36
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.6) | 27.8 (6.2) | 24.8 (3.3) | 26.7 (3.5) | 26.0 (2.2) | 24.8 (3.5) | 26.1 (3.9)
Logical Memory II Subscale, Delayed [Mean (Standard Deviation); unit: units on a scale] — Scores range from 1 to 19; with higher scores indicating better delayed verbal recall.
  units on a scale | 14.2 (3.1) | 13.8 (2.4) | 11.2 (4.0) | 11.3 (3.6) | 13.2 (3.4) | 13.8 (4.4) | 12.9 (3.5)
Clinical Dementia Rating scale (CDR) [Mean (Standard Deviation); unit: units on a scale] — Scores of above 0 indicate progressive decline due to a cognitive disorder.
  units on a scale | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mini Mental State Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 1 to 30; with higher scores indicating better cognitive performance. Scores >25 are normal.
  units on a scale | 29.3 (0.5) | 28.8 (1.5) | 29.5 (0.5) | 29.0 (0.6) | 29.5 (0.8) | 29.5 (0.8) | 29.3 (0.8)
Glasgow Coma Scale (GCS) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 3 to 15; with lower scores indicating impaired consciousness.
  units on a scale | 15.0 (0.0) | 15.0 (0.0) | 15.0 (0.0) | 15.0 (0.0) | 15.0 (0.0) | 15.0 (0.0) | 15.0 (0.0)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 15; with higher scores indicating a greater likelihood of depression.
  units on a scale | 0.0 (0.0) | 0.3 (0.8) | 1.5 (1.5) | 0.8 (1.0) | 1.2 (1.9) | 1.0 (0.9) | 0.8 (1.2)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 30; with higher scores indicating better cognitive performance.
  units on a scale | 28.2 (2.1) | 26.8 (2.3) | 26.5 (3.4) | 26.0 (2.9) | 27.5 (1.4) | 27.2 (1.6) | 27.0 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Count of Treatment Emergent Adverse Events (TEAEs)
Description: A count of participants that experience any adverse events found to be associated with treatment. All adverse events are summarized in the adverse events section.
Time Frame: Up to 7 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 2 | 2 | 1 | 3 | 3

2. Primary Outcome: Count of Lab Abnormalities
Description: Count of participants with clinical lab abnormalities.
Time Frame: Up to 7 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Count of Clinically Significant Changes in Safety Assessments
Description: A count of participants that experienced any clinically significant changes in: Vital Signs, Physical Exam, Electrocardiogram, Neuropsychiatric Inventory - Q, Geriatric Depression Scale, Glasgow Coma Scale, Montreal Cognitive Assessment
Time Frame: Up to 7 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration as determined by pharmacokinetic modeling
Time Frame: Up to 7 days after last dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 21.86 (7.85) | 189.15 (82.18) | 293.22 (150.56) | 125.85 (62.72) | 480.83 (235.19) | 455.65 (167.88)

5. Primary Outcome: Time of Cmax (Tmax)
Description: Time of Cmax as determined by pharmacokinetic modeling
Time Frame: Up to 7 days after last dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.5 (0.548) | 1.67 (0.516) | 2.17 (1.472) | 2.17 (0.983) | 1.83 (0.408) | 3.33 (1.03)

6. Primary Outcome: Area Under the Curve From 0 to 24h (AUC 24h)
Description: Plasma drug exposure as determined by pharmacokinetic modeling, AUC is represented as ng∙h/mL.
Time Frame: Up to 7 days after last dose
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng∙h/mL | 105.29 (48.48) | 993.74 (345.23) | 1547.62 (765.72) | 967.56 (3130.23) | 3130.23 (1655.51) | 3752.1 (1259.84)

7. Secondary Outcome: Receptor Occupancy
Description: Metabotropic glutamate receptor subtype 5 (mGluR5) occupancy using [18F]FPEB Positron Emission Tomography calculated using the percentage of total mGluR5 availability and plasma concentrations of study drug were used to model the relationship between plasma concentration (CP) and receptor occupancy with the conventional sigmoidal maximum receptor occupancy (r_max) model where IC50 is the CP required to produce 50% of the r_max. A nonlinear least squares analysis was used to estimate the parameters from all scans. The data supported a model with 1 parameter (IC50, r_max = 100%). IC80 is the CP required to produce 80% of the r_max. The outcomes of relevance are the IC50 and IC80 calculated for the model.
Time Frame: Up to 24 hours after last dose
Population: Receptor Occupancy is calculated as one value for all participants who underwent [18F]FPEB PET.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- All Participants: Day 1: Admission, administration of study drug, and 2 night in-patient stay; Day 3: Discharge following the completion of all scheduled procedures. . The Receptor Occupancy model is calculated with data from all participants who underwent [18F]FPEB PET.
Arm/Group | All Participants
Number analyzed (Participants) | 8
ng/mL
  IC50 | 33.9 (4)
  IC80 | 136.7 (16)

ADVERSE EVENTS:
Time Frame: Up to 7 days
Arm/Group | 10 mg BMS-984923 | 40 mg BMS-984923 | 70 mg BMS-984923 | 100 mg BMS-984923 | 150 mg BMS-984923 | 200 mg BMS-984923
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 1/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg BMS-984923 (N=6) | 40 mg BMS-984923 (N=6) | 70 mg BMS-984923 (N=6) | 100 mg BMS-984923 (N=6) | 150 mg BMS-984923 (N=6) | 200 mg BMS-984923 (N=6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04805983/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04805983/ICF_001.pdf